CLINICAL TRIAL: NCT06109129
Title: Investıgatıon Of The Effectıveness Of The Mollıı Suıt In Chıldren Wıth Ambulatory Cerebral Palsy: A Double-Blınd Randomızed Controlled Study
Brief Title: Investıgatıon Of The Effectıveness Of The Mollıı Suıt In Chıldren Wıth Ambulatory Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Hidayet Cuha, Lecturer (PHd student), Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023 - 1137
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Spasticity, Muscle
Keywords: Cerebral Palsy; Rehabilitation Technology; Spasticity; Electrotherapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: A Double-Blınd Randomızed Controlled Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessments will be performed by an experienced pediatric physiotherapist blinded to the study hypothesis and design.
  Statistical analysis of the study will be performed by a biostatistician blinded to the study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): First group will participate in the Mollii Suit application for 60 minutes 3 days a week. Mollii Suit consists of a pair of trousers and a jacket. It is a neuromodulation garment consisting of a non-invasive removable control unit that sends electrical signals to the user through electrodes inside. The child will wear the Molli Suit when he/she comes to each session, and the child will be asked to sit or lie down throughout the application in order to avoid any interference with the effectiveness of the suit.
  Interventions: Device: EXOPULSE Mollii Suit
- Control Group (No Intervention): The control group will continue the routine pediatric physiotherapy program 3 days a week. This program, which includes exercises appropriate to the child's motor function level, includes stair climbing, walking exercises, balance, strengthening and flexibility exercises.

INTERVENTIONS:
Device: EXOPULSE Mollii Suit — EXOPULSE Mollii Suit is a personal assistive medical device which is used for low energy whole body transcutaneous electrical stimulation - 20 Volt and 20 Hz. It is composed of a control unit, a jacket and pants with 58 embedded electrodes in direct contact with the skin. EXOPULSE Mollii Suit is used for activation of muscles or relaxation of spastic muscles mediated by a physiological reflex mechanism referred to as reciprocal inhibition. By sending an electrical signal to an antagonistic muscle, the spastic muscle may subsequently relax.
  Arms: Intervention Group

SUMMARY:
Cerebral Palsy (CP) is the most common developmental disorder in childhood. Individuals' independence in daily living activities and participation in education, games, social and community activities are restricted. Technology applications in the field of rehabilitation are gaining momentum. EXOPULSE Mollii Suit method, one of the newest rehabilitation technology products, is a non-invasive neuromodulation approach with a garment that covers the whole body and electrodes placed inside. Designed to improve motor function by reducing spasticity and pain, the method is based on the principle of reciprocal inhibition, which occurs by stimulating the antagonist of a spastic muscle at low frequencies and intensities. Therefore, the aim of our study is to examine the effectiveness of the Mollii Suit application on gross and fine motor function, spasticity severity, balance, walking, selective motor control, postural control, daily living activities, quality of life, pain and sleep quality in individuals with ambulatory spastic CP.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common developmental disorder in childhood and is an umbrella term covering a heterogeneous group of permanent but unchanging movement and posture disorders caused by damage to the developing brain. In a study conducted in Turkey in 2006, the incidence was found to be 4.4 per 1000 live births. While difficulties in selective movement negatively affect motor functions, individuals may also experience difficulties in areas such as communication, behavior, vision, hearing, nutrition, pain and sleep. Individuals' independence in daily living activities and participation in education, games, social and community activities are restricted.

In recent years, the number of systematic reviews and meta-analyses focusing on CP treatments has increased rapidly. These studies are instrumental in providing clinicians and families with newer, safer, and more effective interventions. In a systematic review, it was stated that goal-oriented approaches in the development of gross and fine motor skills prioritize motivation and attention, which are important for neuroplasticity, and that this is necessary for the patient to continue treatment. Rehabilitation technologies such as electrotherapy, virtual reality games, and body weight supported treadmill training, which can be combined with targeted motor training, have been shown to be effective on the patient's gross and fine motor functions.

Technology applications in the field of rehabilitation are gaining momentum. The main reasons for this growth include engineering research, commercial development of rehabilitation products and rapidly growing technological developments. These developments are used in CP rehabilitation to improve motor skills, assist with daily living activities, optimize communication and support academic education.

EXOPULSE Mollii Suit method, one of the newest rehabilitation technology products, is a non-invasive neuromodulation approach with a garment that covers the whole body and electrodes placed inside. Designed to improve motor function by reducing spasticity and pain, the method is based on the principle of reciprocal inhibition, which occurs by stimulating the antagonist of a spastic muscle at low frequencies and intensities. No discomfort or side effects were reported in studies conducted in the pediatric population. In one study, they stated that children felt like superheroes in clothes and that it made them feel good. Families stated that this new approach could be an alternative to current treatments and that it was promising.

In the literature, it has only been applied for the treatment of pain and spasticity in patients with CP, stroke, ataxia and fibromyalgia. Different methodological methods were used in these studies and it was stated that there were inconsistencies between the results. According to a pilot study conducted by Hedin et al., 16 patients with CP at different levels were treated for 60 minutes every other day for 6 weeks, and it was observed that there was a significant decrease in joint range of motion and spasticity severity.

The effectiveness of Mollii Suit on different parameters, especially walking, in individuals with ambulatory CP is unclear and it is stated that better designed studies are needed. Therefore, the aim of our study is to examine the effectiveness of the Mollii Suit application on gross and fine motor function, spasticity severity, balance, walking, selective motor control, postural control, daily living activities, quality of life, pain and sleep quality in individuals with ambulatory spastic CP.

ELIGIBILITY:
Inclusion Criteria:

* Being a voluntary participant in the study,
* Having a diagnosis of spastic CP,
* Being between 1-3 on the Gross Motor Classification System (GMFCS),
* Being between the ages of 4 and 18,
* Being able to express pain and discomfort

Exclusion Criteria:

* Being between 4-5 on Gross Motor Classification System (GMFCS)
* Having Botolunim Toxin A application before 3 months
* Having a surgical intervention before 6 months
* Having a shunt or an invasive medical pump (baclofen, insulin, etc.)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
The Edinburgh Visual Gait Score (EVGS) | 10-15 minutes
  Set up one of the cameras at the end of the 8m walkway track line to capture a coronal view. Place the second camera facing the center of the walkway to capture the sagittal view. The second camera should be set far enough away so as to capture the middle four meters of each trial. A patient should be able to complete two full strides in this distance. Adjust the cameras to be level with the height of the patient's greater trochanter. Record the patient walking back and forth along the walkway. The patient should be barefoot. Open the video recordings in any video player software and take screenshots of each gait cycle event from both coronal and sagittal views. There are 17 observational parameters that should be measured. Each parameter is scored based on either observed condition or measured joint angles. A three-point scale is used for each parameter. After scores have been assigned for each parameter, all scores should be summed.

SECONDARY OUTCOMES:
The Gross Motor Function Measure (GMFM) | 45-60 minutes
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. Items span the spectrum of gross motor activities in five dimensions: lying supine-prone (GMFM-A), sitting (GMFM-B), crawling (GMFM-C), standing (GMFM-D), walking, running and jumping (GMFM-E). GMFM is scored as fourpoint likert between "0" (cannot initiate) and "3" (completed) and calculated as percentage. The score of each section can be used alone or the total score can be calculated. The scale ranging from 0 to 100.
Tardieu Scale | 10-15 minutes
  It is a method that evaluates the velocity-sensitive nature of spasticity through passive movement. Passive stretching is applied slowly (R2) before and fast (R1) after the limb's fall rate against gravity. The difference between R2 and R1 indicates the severity of spasticity. The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle.
Trunk Control Measurement Scale (TCMS) | 15-20 minutes
  The TCMS scale assesses seated trunk control in three dimensions. The maximum score is 58 points where 20 points correspond to static balance, 28 to selective movement control, and 10 to the ability to perform dynamic reaching. The items are scored from 0 to 3, with 0 being the inability to perform the task and 3 being the complete performance of the item. It is an active test where the evaluator gives verbal instructions, demonstrates the movement visually or by guiding the participant, and then asks the participant to perform the test. The best attempt out of three is scored.
Modified Timed Up and Go Test | 3-5 minutes
  Modified TUG is version of TUG test , procedure for TUG test:The TUG test measure is the time taken, in seconds, by an individual to stand up from a standard arm chair, walk a distance of 3 m, turn, walk back to the chair, and sit down again. The subject wears his/her regular footwear. If participants usually use assistive devices such as cane or walker, they should use them during the test, but this should be indicated on the data collection form. No physical assistance is given. Total 3 trial repeats and average time score is recorded.
Modified Functional Reach Test | 3-5 minutes
  Performed with a leveled yardstick that has been mounted on the wall at the height of the patient's acromion level in the non-affected arm while sitting in a chair. Hips, knees and ankles positioned are at 90 degree of flexion, with feet positioned flat on the floor. The initial reach is measured with the patient sitting against the back of the chair with the upper-extremity flexed to 90 degrees, measure was taken from the distal end of the third metacarpal along the yardstick. Consists of three conditions over three trials: Sitting with the back to the wall and leaning right, left and Sitting with the unaffected side near the wall and leaning forward.
Selective Control Assessment of the Lower Extremity (SCALE) | 15 minutes
  The SCALE tool was designed for clinical administrationand scoring by healthcare professionals, to be used in lessthan 15 minutes without specialized equipment. The toolincludes 'Directions for Administration,' 'Instructions forGrading,' and a 'Score Sheet.' Hip, knee, ankle, subtalar,and toe joints are assessed bilaterally. Sitting andside-lying positions allow evaluation of patients who areunable to stand, permit observation of contralateral limbmovements, and enable the patient to visualize their limbin case of proprioceptive deficits. The following factorswere used to develop the assessment and grading criteria:(1) ability to move each joint selectively; (2) involuntarymovement at other joints including the contralateral limb;(3) ability to reciprocate movement; (4) speed of move-ment; and (5) generation of force as demonstrated byexcursion within the available range of motion.
Functional Independence Measure for Children (WeeFIM) | 10-15 minutes
  The WeeFIM consists of 18 items that document functional status. The WeeFIM was scored on a 7-level ordinal scale, ranging from: Independent/No Helper (7-6); Dependent/Helper (5); and Assistance 'Hands On' (4-1) Citation[22]. In addition to a total WeeFIM score, constructed from the sum of 18 independent item scores, there are also three sub-domain scores: Self-care and bowel and bladder management items, mobility and cognition.
The Cerebral Palsy Quality of Life Questionnaire (CP QOL) | 15-20 minutes
  The CP QOL uses a 9- point rating scale to measure how caregivers think their child feels (in general, 1 = very unhappy, 9 = very happy), with scores subsequently being converted to a scale ranging from 0 to 100. The primary caregiver QOL-Child form (children aged 4-12) contains 66 items in seven domains: Social well-being and Acceptance, Functioning, Participation and Physical Health, Emotional Well-being, Pain and Impact of Disability, Access to Services, and Family Health.
Pittsburgh Sleep Quality Index (PSQI) | 10-15 minutes
  PSQI questionnaire assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: Subjective sleep quality, sleep latency, sleep duration, habitual, sleep efficiency, SDs, use of sleeping medication, and daytime dysfunction. Each component score ranges from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range, 0-21). A PSQI global score of ≥5 is considered to be suggestive of significant sleep disorder.
The Wong-Baker Faces Pain Rating Scale | 1-3 minutes
  The Wong-Baker Faces Pain Rating Scale is a method for someone to self-assess and effectively communicate the severity of pain they may be experiencing. The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst."

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Serdaroglu A, Cansu A, Ozkan S, Tezcan S. Prevalence of cerebral palsy in Turkish children between the ages of 2 and 16 years. Dev Med Child Neurol. 2006 Jun;48(6):413-6. doi: 10.1017/S0012162206000910. PMID 16700929
- [Background] Novak I, Hines M, Goldsmith S, Barclay R. Clinical prognostic messages from a systematic review on cerebral palsy. Pediatrics. 2012 Nov;130(5):e1285-312. doi: 10.1542/peds.2012-0924. Epub 2012 Oct 8. PMID 23045562
- [Background] Jones RA, Riethmuller A, Hesketh K, Trezise J, Batterham M, Okely AD. Promoting fundamental movement skill development and physical activity in early childhood settings: a cluster randomized controlled trial. Pediatr Exerc Sci. 2011 Nov;23(4):600-15. doi: 10.1123/pes.23.4.600. PMID 22109783
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Booth ATC, Buizer AI, Meyns P, Oude Lansink ILB, Steenbrink F, van der Krogt MM. The efficacy of functional gait training in children and young adults with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2018 Sep;60(9):866-883. doi: 10.1111/dmcn.13708. Epub 2018 Mar 7. PMID 29512110
- [Background] Chen Y, Fanchiang HD, Howard A. Effectiveness of Virtual Reality in Children With Cerebral Palsy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Jan 1;98(1):63-77. doi: 10.1093/ptj/pzx107. PMID 29088476
- [Background] Salazar AP, Pagnussat AS, Pereira GA, Scopel G, Lukrafka JL. Neuromuscular electrical stimulation to improve gross motor function in children with cerebral palsy: a meta-analysis. Braz J Phys Ther. 2019 Sep-Oct;23(5):378-386. doi: 10.1016/j.bjpt.2019.01.006. Epub 2019 Jan 23. PMID 30712812
- [Background] van Hedel HJA, Severini G, Scarton A, O'Brien A, Reed T, Gaebler-Spira D, Egan T, Meyer-Heim A, Graser J, Chua K, Zutter D, Schweinfurther R, Moller JC, Paredes LP, Esquenazi A, Berweck S, Schroeder S, Warken B, Chan A, Devers A, Petioky J, Paik NJ, Kim WS, Bonato P, Boninger M; ARTIC network. Advanced Robotic Therapy Integrated Centers (ARTIC): an international collaboration facilitating the application of rehabilitation technologies. J Neuroeng Rehabil. 2018 Apr 6;15(1):30. doi: 10.1186/s12984-018-0366-y. PMID 29625628
- [Background] Pennati GV, Bergling H, Carment L, Borg J, Lindberg PG, Palmcrantz S. Effects of 60 Min Electrostimulation With the EXOPULSE Mollii Suit on Objective Signs of Spasticity. Front Neurol. 2021 Oct 15;12:706610. doi: 10.3389/fneur.2021.706610. eCollection 2021. PMID 34721255
- [Background] Arkkukangas M, Hedberg Graff J, Denison E. Evaluation of the electro-dress Mollii® to affect spasticity and motor function in children with cerebral palsy: Seven experimental single-case studies with an ABAB design. 2022;9(1). doi:10.1080/23311916.2022.2064587
- [Background] Hedin H, Wong C, Sjödén A. The effects of using an electrodress (Mollii®) to reduce spasticity and enhance functioning in children with cerebral palsy: a pilot study. https://doi.org/101080/2167916920201807602. 2020;24(3):134-143. doi:10.1080/21679169.2020.1807602
- [Background] Jonasson LL, Sorbo A, Ertzgaard P, Sandsjo L. Patients' Experiences of Self-Administered Electrotherapy for Spasticity in Stroke and Cerebral Palsy: A Qualitative Study. J Rehabil Med. 2022 Feb 14;54:jrm00263. doi: 10.2340/jrm.v53.1131. PMID 34935050
- [Background] Nordstrom B, Prellwitz M. A pilot study of children and parents experiences of the use of a new assistive device, the electro suit Mollii. Assist Technol. 2021 Sep 3;33(5):238-245. doi: 10.1080/10400435.2019.1579267. Epub 2019 Apr 4. PMID 30945989
- [Background] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Background] Rubio-Zarapuz A, Apolo-Arenas MD, Clemente-Suarez VJ, Costa AR, Pardo-Caballero D, Parraca JA. Acute Effects of a Session with The EXOPULSE Mollii Suit in a Fibromyalgia Patient: A Case Report. Int J Environ Res Public Health. 2023 Jan 26;20(3):2209. doi: 10.3390/ijerph20032209. PMID 36767576
- [Background] Arkkukangas M, Graff JH, Denison E. Evaluation of the electro-dress Mollii® to affect spasticity and motor function in children with cerebral palsy: Seven experimental single-case studies with an ABAB design. Cogent Eng. 2022;9. doi:10.1080/23311916.2022.2064587
- [Background] Russell DJ, Avery LM, Rosenbaum PL, Raina PS, Walter SD, Palisano RJ. Improved scaling of the gross motor function measure for children with cerebral palsy: evidence of reliability and validity. Phys Ther. 2000 Sep;80(9):873-85. PMID 10960935
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Boyd RN, Kerr Graham H. Objective measurement of clinical findings in the use of botulinum toxin type A for the management of children with cerebral palsy. Europenn Journul qf Neurology. 1999;6:23-35. doi:10.1111/j.1468-1331.1999.tb00031.x
- [Background] Numanoglu A, Gunel MK. Intraobserver reliability of modified Ashworth scale and modified Tardieu scale in the assessment of spasticity in children with cerebral palsy. Acta Orthop Traumatol Turc. 2012;46(3):196-200. doi: 10.3944/aott.2012.2697. PMID 22659636
- [Background] Heyrman L, Molenaers G, Desloovere K, Verheyden G, De Cat J, Monbaliu E, Feys H. A clinical tool to measure trunk control in children with cerebral palsy: the Trunk Control Measurement Scale. Res Dev Disabil. 2011 Nov-Dec;32(6):2624-35. doi: 10.1016/j.ridd.2011.06.012. Epub 2011 Jul 14. PMID 21757321
- [Background] Ozal C, Ari G, Gunel MK. Inter-intra observer reliability and validity of the Turkish version of Trunk Control Measurement Scale in children with cerebral palsy. Acta Orthop Traumatol Turc. 2019 Sep;53(5):381-384. doi: 10.1016/j.aott.2019.04.013. Epub 2019 Jul 11. PMID 31303422
- [Background] Dhote SN, Khatri PA, Ganvir SS. Reliability of "Modified timed up and go" test in children with cerebral palsy. J Pediatr Neurosci. 2012 May;7(2):96-100. doi: 10.4103/1817-1745.102564. PMID 23248683
- [Background] Bartlett D, Birmingham T. Validity and reliability of a pediatric reach test. Pediatr Phys Ther. 2003 Summer;15(2):84-92. doi: 10.1097/01.PEP.0000067885.63909.5C. PMID 17057438
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Ong AM, Hillman SJ, Robb JE. Reliability and validity of the Edinburgh Visual Gait Score for cerebral palsy when used by inexperienced observers. Gait Posture. 2008 Aug;28(2):323-6. doi: 10.1016/j.gaitpost.2008.01.008. Epub 2008 Mar 6. PMID 18328710
- [Background] Rathinam C, Bateman A, Peirson J, Skinner J. Observational gait assessment tools in paediatrics--a systematic review. Gait Posture. 2014 Jun;40(2):279-85. doi: 10.1016/j.gaitpost.2014.04.187. Epub 2014 Apr 18. PMID 24798609
- [Background] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Background] James S, Ziviani J, Boyd R. A systematic review of activities of daily living measures for children and adolescents with cerebral palsy. Dev Med Child Neurol. 2014 Mar;56(3):233-44. doi: 10.1111/dmcn.12226. Epub 2013 Aug 13. PMID 23937056
- [Background] Atasavun Uysal S, Duger T, Elbasan B, Karabulut E, Toylan I. Reliability and Validity of The Cerebral Palsy Quality of Life Questionnaire in The Turkish Population. Percept Mot Skills. 2016 Feb;122(1):150-64. doi: 10.1177/0031512515625388. Epub 2016 Feb 1. PMID 27420313
- [Background] Miro J, Castarlenas E, de la Vega R, Sole E, Tome-Pires C, Jensen MP, Engel JM, Racine M. Validity of three rating scales for measuring pain intensity in youths with physical disabilities. Eur J Pain. 2016 Jan;20(1):130-7. doi: 10.1002/ejp.704. Epub 2015 Mar 31. PMID 25833415
- [Background] Kingsnorth S, Orava T, Provvidenza C, Adler E, Ami N, Gresley-Jones T, Mankad D, Slonim N, Fay L, Joachimides N, Hoffman A, Hung R, Fehlings D. Chronic Pain Assessment Tools for Cerebral Palsy: A Systematic Review. Pediatrics. 2015 Oct;136(4):e947-60. doi: 10.1542/peds.2015-0273. PMID 26416940
- [Background] Bakir E. Pediatric Pain Assessment and Tools: The Influence of Culture and Age on Pain Assessment. Published online 2017. doi:10.5336/nurses.2016-52467
- [Background] Erwin AM, Bashore L. Subjective Sleep Measures in Children: Self-Report. Front Pediatr. 2017 Feb 13;5:22. doi: 10.3389/fped.2017.00022. eCollection 2017. PMID 28243584
- [Result] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477